CLINICAL TRIAL: NCT07268417
Title: Group Medical Appointments for Intensive Lifestyle Treatment for Obesity in Cleveland Clinic Primary Care Practices
Acronym: ACTIVATE OC
Status: Enrolling by invitation | Type: Observational
Sponsor: Anita Misra-Hebert (Other)
Collaborators: Patient-Centered Outcomes Research Institute (Other); The Cleveland Clinic (Other)
Responsible Party: Sponsor-Investigator, Anita Misra-Hebert, Professor of Medicine, Cleveland Clinic Lerner College of Medicine of Case Western Reserve University; Staff, Department of Internal Medicine; Director, Healthcare Delivery and Implementation Science Center, The Cleveland Clinic
Organization: The Cleveland Clinic (Other)
Other Study IDs: 24-1147; PCORI Funded (Other: Patient-Centered Outcomes Research Institute)
Record Dates: First submitted 2025-11-13; First posted 2025-12-05 (Actual); Last update posted 2026-01-09 (Actual); Status verified 2025-11

CONDITIONS: Obesity & Overweight
Keywords: Shared Medical Appointment Obesity Care; Intensive Lifestyle Treatment for Obesity; ACTIVATE OC
MeSH Terms: conditions — Obesity; Overweight

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Other
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: ACTIVATE OC — Offering of Shared Medical Appointments for Obesity Treatment

SUMMARY:
In 2023, Cleveland Clinic was accepted into a national program, the Patient-Centered Outcomes Research Institute Health Systems Implementation Initiative (PCORI HSII) which aims to improve implementation of prior published PCORI-funded research evidence into real-world practice. The investigators first received funding to build organizational capacity to participate in health system implementation projects. This protocol describes activities for our first implementation project for which the investigators have received funding from the PCORI HSII program.

The investigator's project seeks to expand the availability of shared medical appointments (SMAs) for obesity treatment in all 56 primary care practices of the Cleveland Clinic health system in Northeast Ohio. The proposed project, to be implemented as part of routine healthcare delivery, will adapt aspects of a prior study funded by the PCORI that generated evidence that group visits such as SMAs can help with obesity treatment. All primary care patients in Northeast Ohio with obesity (body mass index (BMI) >/=30) and aged between 20 and 75 years will be potentially eligible for enrollment in the SMAs. Primary care providers will offer patients entry into the SMAs as part of usual clinical care during office visits. In addition, information about these SMAs will also be available to the patients through the "MyChart" patient portal in EPIC. Implementation of the SMAs will happen in three phases (pre-implementation, active implementation, and maintenance) over 42 months. During its implementation, the project intends to reach over 140,000 patients. Quantitative and qualitative methods will be used to evaluate implementation and effectiveness outcomes associated with the SMAs. Electronic medical records and patient surveys will be the key data sources for the quantitative evaluation. Qualitative data collection methods will include semi-structured interviews, field observations, and periodic reflections.

As this implementation project will be part of routine care delivery, the investigators emphasize that the risks (physical, psychological, social, legal, financial, or other) associated with participation in SMAs for obesity will not be greater than minimal or those posed by any SMAs as currently configured for the delivery of other healthcare services within the Cleveland Clinic healthcare system. The potential benefits associated with participation in these SMAs include weight loss, improvements in cardiovascular risk factors, and reduced utilization of acute healthcare services.

DETAILED DESCRIPTION:
The objective of this implementation effort is to optimize the availability of intensive lifestyle treatment of obesity in the adult population of patients who receive care within the Cleveland Clinic health system in Northeast Ohio primary care practices as part of routine clinical practice. Utilizing the group visit model from the evidence generated from the Befort et al Patient-Centered Outcomes Research (PCORI) funded study,(5) the investigators will significantly expand current health system obesity treatment resources and build on our model of SMAs led by multidisciplinary teams to deliver the intervention. Through a coordinated health system-wide implementation effort in all primary care practices, the investigators aim to improve the health of our patients with obesity through developing a successful obesity treatment program, improving upon current health system programs, with the goal of long-term impact in reducing patient comorbidities, cardiovascular risk, and promoting sustainable weight loss. The investigators propose to implement group visits for intensive lifestyle intervention for obesity utilizing the SMA model. Implementation of the Obesity SMAs will be in all 56 Cleveland Clinic primary care practices in Northeast Ohio.

Specific Aims

Aim 1. To prepare for implementation of Obesity Treatment SMAs across all Northeast Ohio Primary Care Practices (Pre-Implementation)

Pre-Implementation Phase (9 months)

* Adaptation of Obesity SMA Training Materials for Primary Care Providers with input from Continuous Improvement Specialists regarding practice change principles
* Delivery of Education Sessions, including topic of implementation outcomes
* Quantitative Assessment of Practice Variation in Obesity Treatment Patterns
* Qualitative Assessment of Barriers and Facilitators to Obesity Treatment at Primary Care Practice Level
* Creation of Clinical Decision Support Tool for SMA referral
* Creation of Patient and Employee Advisory Panel

Aim 2. To Implement Obesity Treatment SMAs across all Northeast Ohio Primary Care Practices (Active Implementation)

Active Implementation Phase (18 months)

* Implementation of Clinical Decision Support at Implementation Sites
* Delivery of Additional Educational Materials to Implementation Sites to refresh learning
* Practice Facilitation at Implementation Sites
* Delivery of Obesity SMA Intervention
* Qualitative and Survey Data Collection regarding- Patient and Provider Implementation Outcomes of acceptability, feasibility, appropriateness
* Quantitative Data Collection of Implementation Outcomes of adoption, fidelity, effectiveness, implementation cost
* Patient and Employee Advisory Panel Input into Implementation Evaluation

Aim 3: To monitor and evaluate the maintenance of the Obesity Treatment SMAs across all Northeast Ohio Primary Care Practices (Maintenance & Sustainment)

Maintenance & Sustainment Phase (15 months)

* Quantitative Data Collection of Implementation Outcomes- adoption, fidelity, effectiveness, cost- with comparison to active implementation phase
* Capture Practice Level adaptations with comparison to active implementation phase.

Study Population (Potential Eligible / Intended Reach) Potentially eligible patients: Utilizing electronic medical record data, the investigators determined across the 56 outpatient primary care practices, the total patient population ages 20-75 with a body mass index (BMI) >/= 30 who have had a primary care visit within the past 18 months is 170,087 patients.

Intended reach: The intended reach will exclude patients with a history of bariatric surgery, current pregnancy, current cancer diagnosis or cognitive impairment diagnosis. Exclusion criteria are based upon unique clinical situations affecting BMI as well as conditions that may affect SMA participation. Prior obesity SMA participation will not be an exclusion. The intended reach includes 141,735 potentially eligible patients ages 20 to 75, with an office visit within 18 months, BMI >/=30, with exclusion of history of bariatric surgery, pregnancy, current cancer diagnosis or cognitive impairment diagnosis. Through navigator support, the investigators will assess demographic distribution of patients with uptake of the program and will ensure representation from groups with higher Area Deprivation Index (ADI). If this is not the case, the investigators will conduct outreach to eligible patients outside of an office visit, through the MyChart portal or telephone outreach. Scripts will be created as part of routine clinical care during the pre-implementation phase.

Entry Into SMAs Entry into the obesity treatment program will be offered by a patient's primary care provider as part of usual clinical care and can be offered at the time of an office visit. In addition, the clinical and project teams will create flyers describing the program to be available to primary care practices. This information will also be available through our MyChart patient portal in the EPIC(6) electronic medical record. Scripts will be created as part of routine clinical care during the pre-implementation phase.

Once the referral to the program is made, the patient will complete an individual appointment, offered as both in-person or virtual, with either an obesity-trained primary care provider, an endocrinology provider, or a Wellness Medicine provider from the Primary Care Institute. This individual appointment will be focused on discussion of the diagnosis of obesity and treatment options, including the SMA program. If the patient accepts the referral to the SMA, the first appointment will be scheduled. The program will include options of scheduling both the initial individual appointment and the SMA through the primary care practice office or an opportunity for self-scheduling through our MyChart patient portal. Throughout the study, the investigators will have primary care navigator support to ensure outreach to underrepresented groups.

ELIGIBILITY:
Inclusion Criteria:

* patient population ages 20-75 with a body mass index (BMI) >/= 30 who have had a primary care visit within the past 18 months

Exclusion Criteria:

* history of bariatric surgery, pregnancy, current cancer diagnosis or cognitive impairment diagnosis

Ages: 20 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients who see a primary care provider within one of the Cleveland Clinic Health System Northeast Ohio 56 primary care sites, that meet the inclusion/exclusion criteria.
Sampling Method: Non-Probability Sample
Enrollment: 3600 (Estimated)
Dates: Start 2024-12-01 (Actual); Primary Completion 2028-02 (Estimated); Study Completion 2028-05 (Estimated)

PRIMARY OUTCOMES:
Weight Loss | Measured at baseline, every 6 months during the intervention, and 6 months post-intervention.
  Change in body weight as measured in kg compared to baseline weight.

SECONDARY OUTCOMES:
Weight Loss | Baseline, every 6 months during intervention, and 6 months post-intervention
  Change in body weight as measured in a percentage of total weight compared to baseline.
Outcome measure type: Reach | Timing and frequency of measurement is every 3 months.
  Actual reach measuring the overall total number of patients:
  * Program participation (offered): total number of patients who are offered the program.
  * Program participation (enrolled): total number of patients who are enrolled in the program.
  * Program participation (completed): total number of patients who complete the program.
Outcome measure type: Effectiveness | Hospitalizations and emergency department visits - every 6 months
  Hospitalizations and emergency department visits: number of acute care hospitalizations, number of emergency department visits. Determining association between obesity treatment and acute care utilization.
Outcome measure type: Effectiveness | Baseline and end of intervention
  Body Composition (body impedance analysis machine): subset of patients electing to have measurement
Patient Reported Outcomes- PROMIS10 Global Health Survey | Baseline, every month during the SMA intervention and 6 months post-intervention.
  PROMIS-10 Global Health (8) instrument routinely collected from Cleveland Clinic patients and utilized in Endocrinology SMAs as part of Obesity Survey to assess change in item scores over time.
Provider Bias Related to Patients with Obesity survey | Administered at baseline and at end of intervention period.
  Fat Phobia Scale-14 Item Short Form survey to assess primary care providers change in bias item scores over time.
Provider views of Acceptability, Appropriateness, Feasibility survey | Administered to primary care providers every 6 months starting baseline throughout active implementation & maintenance.
  Captured through surveys, provider views of Acceptability, Appropriateness, Feasibility (19). Providers views of intervention may impact adoption of intervention for patients. Measured by change in item scores over time.
Outcome Measure: Adoption (Actual) | Every 3 months during the intervention period
  Number of primary care providers in each practice group referring to obesity SMA will be measured by number of referrals attributed to practice group.
Outcome measure: SMA Leader Adoption | Every 3 months during intervention period.
  Number of obesity trained providers who are trained to lead SMAs who participate in program as SMA leader measured by number of SMAs attributed to eligible providers.
Formal Qualitative Assessment of context of high referral and low referral practices: Pre-implementation | Pre-implementation
  To understand barriers and facilitators to uptake of obesity treatment
  * Semi-structured interviews with non-patient (employee) key stakeholders at high/low referral sites
  * Direct field observations of high/low referral practice sites Qualitative methodologists will analyze the qualitative data (transcripts and descriptive fieldnotes) will be coded to reflect key domains of interest and emergent themes. Demographics of the qualitative sample will be reported in aggregate.
Formal Qualitative Assessment: Observations of Employee and Patient Advisory Panels | Quarterly meetings throughout pre- and active implementation.
  To examine anticipated barriers and facilitators to implementation and to assess ongoing implementation activities. Qualitative methodologists will analyze the qualitative data (fieldnotes) will be coded to reflect key domains of interest and emergent themes.
Formal Qualitative Assessment: Semi-structured Interviews with Patients at High/Low Referral Sites | Baseline, 6 months, 12 months during active implementation
  Inviting a sample of patients receiving the intervention at high and low referral sites to participate in interviews to assess perceptions of acceptability of and satisfaction with group visits for intensive lifestyle intervention for obesity. Qualitative methodologists will analyze the qualitative data (transcripts) will be coded to reflect key domains of interest and emergent themes. Demographics of the qualitative sample will be reported in aggregate.
Formal Qualitative Assessment: Periodic Reflections with Agents of Implementation | Monthly or bimonthly throughout active implementation and maintenance.
  Periodic reflections conducted with a subgroup of pool of obesity trained providers and weight management navigators across practice locations to understand barriers and facilitators to uptake of obesity treatment.
  Qualitative methodologists will analyze the qualitative data (descriptive fieldnotes) will be coded to reflect key domains of interest and emergent themes.
Outcome measure type: Effectiveness | Every 6 months
  Outpatient visits: number of outpatient visits (in clinic or virtual, primary care and specialty). Determining association between obesity treatment and outpatient utilization.
Outcome measure type: Effectiveness | Baseline, every 6 months during intervention, and 6 months post-intervention
  Glycosylated Hemoglobin: change in A1c as measured in a percentage compared to baseline to assess effect of obesity treatment on glycemic control.
Outcome measure type: Effectiveness | Baseline, every 6 months during intervention, and 6 months post-intervention
  Low Density Lipoprotein (LDL) Triglycerides measured in mg/dl compared to baseline to assess effect of obesity treatment on lipid control.
Outcome measure type: Effectiveness | Baseline, every 6 months during intervention, and 6 months post-intervention
  Blood pressure as measured in mmHg to assess effect of obesity treatment on blood pressure control.
Patient Reported Outcomes - Obesity history, diabetes/hypoglycemia history if relevant, diet, exercise Survey | Baseline, then follow-up survey every month during AMS intervention.
  Surveys currently utilized in Department of Endocrinology SMAs to assess change in item scores over time.
Outcome Measure: Adoption (Actual) | Every 3 months during intervention period
  Number of primary care providers in each practice group referring to obesity SMA will be measured by the percentage of referrals attributed to practice group.
Outcome Measure: SMA Leader Adoption | Every 3 months during intervention period
  Percentage of obesity trained providers who are trained to lead SMA who participate in program as an SMA leader will be measured by percentage of SMAs attributed to eligible providers.
Outcome measure type: Reach (Other) | At 18 months post intervention start time of Practice Group 1, then every 3 months until end of study.
  (Other) reach - * Session attendance rate: proportion of sessions attended per person (average and distribution) measured by percentage of sessions completed.

CONTACTS AND LOCATIONS:
Locations (1):
- Cleveland Clinic, Cleveland, Ohio, United States

IPD SHARING:
Plan to Share IPD: No
Data used for this study will include human research participant data that are sensitive and cannot be publicly shared due to legal and ethical restrictions by the Cleveland Clinic regulatory bodies, including the institutional review board and legal counsel. We will make our data sets available on request, under appropriate data use agreements with the specific parties interested in academic collaboration.

REFERENCES:
- [Background] Bacon JG, Scheltema KE, Robinson BE. Fat phobia scale revisited: the short form. Int J Obes Relat Metab Disord. 2001 Feb;25(2):252-7. doi: 10.1038/sj.ijo.0801537. PMID 11410828
- [Background] Hays RD, Bjorner JB, Revicki DA, Spritzer KL, Cella D. Development of physical and mental health summary scores from the patient-reported outcomes measurement information system (PROMIS) global items. Qual Life Res. 2009 Sep;18(7):873-80. doi: 10.1007/s11136-009-9496-9. Epub 2009 Jun 19. PMID 19543809
- [Background] Weiner BJ, Lewis CC, Stanick C, Powell BJ, Dorsey CN, Clary AS, Boynton MH, Halko H. Psychometric assessment of three newly developed implementation outcome measures. Implement Sci. 2017 Aug 29;12(1):108. doi: 10.1186/s13012-017-0635-3. PMID 28851459
- [Background] Befort CA, VanWormer JJ, Desouza C, Ellerbeck EF, Gajewski B, Kimminau KS, Greiner KA, Perri MG, Brown AR, Pathak RD, Huang TT, Eiland L, Drincic A. Effect of Behavioral Therapy With In-Clinic or Telephone Group Visits vs In-Clinic Individual Visits on Weight Loss Among Patients With Obesity in Rural Clinical Practice: A Randomized Clinical Trial. JAMA. 2021 Jan 26;325(4):363-372. doi: 10.1001/jama.2020.25855. PMID 33496775